CLINICAL TRIAL: NCT05903794
Title: An Open-label, Dose-escalation Study to Evaluate the Safety and Tolerability of Gene Therapy With EXG102-031 in Participants With Neovascular Age-related Macular Degeneration.
Brief Title: A Study of EXG102-031 in Patients With wAMD (Everest)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exegenesis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG102-031 (211)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration (nAMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Dose-escalation Study with four cohorts of three participants in each.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXG102-031 (Experimental): Each participant will receive a single subretinal injection of EXG102-031 in the study eye. Participants will be enrolled into one of four dosage groups sequentially, and the dose administered will be determined based on which study group the participant is enrolled into.
  Interventions: Biological: EXG102-031

INTERVENTIONS:
Biological: EXG102-031 — EXG102-031 is a recombinant adeno-associated virus (rAAV) expressing an angiopoietin domain and VEGF receptor (ABD-VEGFR) fusion protein. EXG102-031 will be administered by subretinal injecting into one eye of each participant.

SUMMARY:
In neovascular (wet) age-related macular degeneration (nAMD), the macula, or the part of the eye that provides the clear, detailed central vision, is being affected by abnormal blood vessel growth and leakage. This leakage affects the vision over time and can lead to severe blurriness or blinding. EXG102-031 was made to block the extra vessel formation which would lead to less leakage affecting the vision. Before EXG102-031 can be tested for its efficacy (if it makes vision better), it must be tested to see if it is safely tolerated to confirm it can continue to be studied in more patients with nAMD.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a major cause of blindness and visual impairment in older adults. The wet form of AMD, also called neovascular AMD (nAMD) usually causes faster vision loss than the dry form. The most common current treatments of nAMD are products that inhibit vascular endothelial growth factor (VEGF) (including ranibizumab (LUCENTIS®, Genentech) and aflibercept (EYLEA®, Regeneron) and are delivered by intravitreal injections at 4 to 16 week intervals and continued indefinitely. This Phase I, open-label, multiple-cohort, dose-escalation study is designed to evaluate the safety and tolerability of EXG102-031 gene therapy in subjects with previously treated nAMD. Safety will be assessed over 52 weeks after the administration of EXG102-031.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 50 years of age;
2. Diagnosis of nAMD and current active lesion in the study eye at Screening;
3. An ETDRS BCVA letter scores between 73 and 19 letters in the study eye;
4. Response to anti-VEGF treatment during Screening;
5. The study eye must be a pseudophakic lens (post-cataract surgery status); and
6. Voluntarily agree to participate in the clinical trial, understand the trial procedures, and be capable of signing the informed consent form before screening.

Exclusion Criteria:

1. Presence of any ocular disease or history of disease in the study eye other than nAMD that may affect central visual acuity and/or macular detection, including retinal detachment, or in the opinion of the investigator could limit VA improvement in the study eye;
2. Presence in the study eye of CNV or macular edema due to causes other than AMD;
3. Presence in the study eye of scarring, fibrosis or atrophy involving the macula;
4. Subretinal hemorrhage accumulating in the center of the macula of the test eye, with an area of hemorrhage ≥ 4 optic disc diameters;
5. Active ocular infection in either eye;
6. Presence of advanced glaucoma or uncontrolled glaucoma in the study eye;
7. History of intraocular surgery in the study eye within 90 days of screening; or
8. Prior receipt of any ocular or systemic gene therapy agent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability | Throughout 52 weeks
  Frequency, type, and intensity of ocular and non-ocular adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Evaluation of potential efficacy | 52 weeks post administration
  Change from baseline in best corrected visual acuity (BCVA) measured by ETDRS method
Evaluation of potential safety | Through week 24
  Frequency, type, and intensity of ocular and non-ocular adverse events (AEs) and serious adverse events (SAEs)
Evaluation of supplementary therapy injections received | Throughout 52 weeks post administration
  Average number of doses of anti-vascular endothelial growth factor (VEGF) supplemental therapy received

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Khanani, MD, Principal Investigator — Sierra Eye Associates
Locations (2):
- United States (2):
  - Sierra Eye Associates, Reno, Nevada
  - Erie Retina Research, Erie, Pennsylvania

IPD SHARING:
Plan to Share IPD: No